CLINICAL TRIAL: NCT06039709
Title: Pilot Study of Sonodynamic Therapy With 5-ALA for the Treatment of Recurrent Glioblastoma Using Neuronavigation-Guided Low-Intensity Focused Ultrasound
Brief Title: Sonodynamic Therapy in Patients With Recurrent GBM
Acronym: GBM 001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shayan Moosa, MD (Other)
Responsible Party: Sponsor-Investigator, Shayan Moosa, MD, Assistant Professor of Neurosurgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR230064
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Glioblastoma; Glioblastoma Multiforme; GBM
Keywords: Sonodynamic Therapy; Low-Intensity Focused Ultrasound (LIFU); Focused Ultrasound; 5-ALA; Brain Cancer
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Sonodynamic Therapy (5-ALA + LIFU) (Experimental): Administration of SDT occurs 1-3 weeks prior to GBM resection
  Interventions: Combination Product: 5-ALA and Low-Intensity Focused Ultrasound (SDT)

INTERVENTIONS:
Combination Product: 5-ALA and Low-Intensity Focused Ultrasound (SDT) — 5-ALA (20mg/kg orally) given ~6 hours prior to LIFU. Focused ultrasound will target a maximum of 50% of the tumor.

SUMMARY:
Patients diagnosed with glioblastoma (GBM) are faced with limited treatment options. This pilot study will evaluate the safety and feasibility of combining an investigational drug called 5-ALA with neuronavigation-guided low-intensity focused ultrasound (LIFU) for patients who have recurrent GBM. Focused ultrasound (FUS) can be used to non-invasively destroy tumor tissue while preserving normal tissue. When FUS is combined with 5-ALA, this combinatorial approach is called sonodynamic therapy (SDT), and this investigational therapy is being tested for its ability to cause damage to GBM cells. SDT will take place prior to surgery for recurrent GBM.

DETAILED DESCRIPTION:
The combination of 5-ALA (Gleolan) and LIFU is collectively known as sonodynamic therapy (SDT). SDT is an investigational therapy that will be administered 1-3 weeks before surgery for recurrent GBM. Researchers seek to determine the safety and feasibility of this therapy as well as measure its effectiveness to elicit tumor-cell death. All participants are expected to stay overnight in the hospital following administration of SDT to monitor for adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Disease status and Disease Parameters:

   * Suspected recurrent glioblastoma that is clearly measurable based on the modified Response Assessment in Neuro-Oncology (RANO) criteria
   * The tumor lesion needs to comprise at least 1 contrast-enhancing lesion with a volume of ≥ 2 cm3 and ≤ 20 cm3 of targeted treatment area
   * Tumor tissue to be treated is in a surgically accessible brain region for resection
   * The brain tumor to be treated must be in the treatment envelope of the NaviFUS system (30 mm to 90 mm from the inner skull table)
   * Recurrence will be assessed by imaging and confirmed by consensus at tumor board
2. Men or women between the ages of 18-80 years of age at the time of consent
3. No contraindication to repeat brain surgery
4. Karnofsky Performance Score of 70-100
5. Able to undergo an MRI with contrast
6. Able to swallow oral medications
7. Willingness and ability to comply with scheduled visits, treatment plans, lifestyle considerations, laboratory tests, and other procedures.
8. Ability to understand and the willingness to sign a written informed consent document (personally or by the legally authorized representative, if applicable).
9. Participants who received prior chemotherapy, radiation therapy, immunotherapy, and/or another investigational therapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1 or baseline) from the acute effects of the therapy or therapies) except for residual alopecia or Grade 2 peripheral neuropathy prior to registration.
10. Has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by the local laboratory for eligibility):

Hematological

* Absolute neutrophil count (ANC) ≥1000/mm3
* Platelets ≥ 100,000/mm3
* Hemoglobin ≥ 11 g/dL for women and ≥ 12 g/dL for men Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator.
* INR ≤ 1.4

Renal & Hepatic

* Creatinine clearance CrCl ≥ 60 mL/min/1.73 m2 as estimated by the Cockcroft-Gault (C-G) equation. If estimated CrCl is abnormal, accurate measurement should be obtained by 24- hour CrCl.
* Bilirubin ≤ 1.5 x ULN (except in patients with Gilbert's disease, where bilirubin to 2.0x ULN is allowed).
* AST and ALT ≤ 3 x ULN
* Alkaline phosphatase ≤ 3 x ULN
* Estimated glomerular filtration rate ≥30mL/min/1.73m2

Exclusion Criteria:

1. Known sensitivity or allergy to 5-ALA
2. Simultaneous use of other potentially phototoxic substances (e.g. tetracyclines, sulfonamides, fluoroquinolones, hypericin extracts)
3. Diagnosis of porphyria
4. Hypersensitivity against porphyrins
5. Pregnancy
6. Significant cardiac disease or coagulopathy
7. Herniation / intractable seizure / other clinical indications requiring urgent resection
8. Known active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C (for example, hepatitis B surface antigen positive)
9. Have had a recent (≤3 months prior to registration) transient ischemic attack or stroke
10. Significant vascular disease (e.g. aortic aneurysm)
11. Evidence of bleeding diathesis or coagulopathy
12. Need for systemic anticoagulation which cannot be held for 7 days prior to SDT
13. Unstable angina and/or congestive heart failure (NYH Class III or Class IV; see section 13.2) within 6 months prior to registration
14. Severe hypertension (systolic ≥ 180 mm Hg; diastolic ≥ 120 mm Hg) despite anti-hypertensive medications
15. Transmural myocardial infarction within 6 months prior to registration
16. Serious and inadequately controlled cardiac arrhythmia
17. Acute exacerbation of chronic obstructive pulmonary disease
18. Has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study
19. Treatment with another investigational drug or investigational procedure within 30 days prior to registration or within 5 half-lives of the investigational product, whichever is longer
20. Brain edema and/or mass effect that causes midline shift of more than 15 mm
21. Evidence of recent (within 30 days prior to registration) intracranial hemorrhage
22. Calcifications or metallic implanted objects in the focused ultrasound sonication path
23. Scalp atrophy or scars at the expected location of transducer
24. Cerebral or systemic vasculopathy
25. Need for or currently on dialysis
26. Respiratory: chronic pulmonary disorders (e.g., severe emphysema, COPD, pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area).
27. Receipt of radiotherapy ≤21 days prior to registration
28. Receipt of chemotherapy ≤ 21 days prior to registration
29. Prior treatment with sonodynamic therapy
30. Concurrent use of Optune device
31. Concurrent use of supplements or medications with substantial antioxidant effects (including sulfhydryl-containing medications such as captopril or supplements such as N-acetylcysteine, or high doses of vitamins with antioxidant activity such as C or E)
32. Known sensitivity to gadolinium

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From informed consent through 30 days after study intervention is complete
  Per NCI Common Terminology Criteria for Adverse Events v5.0
Severity of adverse events | From informed consent through 30 days after study intervention is complete
  Per NCI Common Terminology Criteria for Adverse Events v5.0
Incidence of intracranial hemorrhage and/or worsening of edema | From day after SDT (day 1) up to the time of surgery (day 7-day 21)
  On post-SDT MRIs
Extent of targeted tumor area receiving FUS | Day 0
  Use of NaviFUS system to target a maximum of 50% of the tumor volume of one contiguous lesion
Ability to have participants undergo planned surgery without delay | within 3 weeks following SDT
  A delay is defined as more than 3 weeks after SDT

SECONDARY OUTCOMES:
Response of target tissue following SDT on imaging | From day after SDT (day 1) up to 100 days after intervention is completed
  Via MRI w/ use of modified Response Assessment in Neuro-Oncology (RANO) criteria
Histologic tumor devitalization | Day 7-Day 21
  Evaluating cell fate and cell death via histologic samples after GBM resection

CONTACTS AND LOCATIONS:
Overall Officials: Shayan Moosa, MD, Principal Investigator — UVA
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No